CLINICAL TRIAL: NCT00027105
Title: Morbidity Following the Diagnosis and Treatment of Patients With Breast Cancer: A Multi-Institutional Study Between the National Institutes of Health (NIH) Rehabilitation Medicine Department (RMD) and the Walter Reed National Military Medical Center (WRNMMC) Breast Care Center
Brief Title: Morbidity Following the Diagnosis and Treatment of Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 020044; 02-CC-0044; NCT00514176 (obsolete NCT alias)
Record Dates: First submitted 2001-11-20; First posted 2001-11-21 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-08-17

CONDITIONS: Breast Cancer; Lymphedema; Physical Therapy; Shoulder
Keywords: Fatigue; Shoulder function; Lymphedema; Breast Cancer; Breast Cancer Surgery; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine the frequency and severity of problems in women with breast cancer during the first year after initial medical treatment, including:

* Physical impairments, such as loss of strength or flexibility, increased weight and swelling
* Symptom distress, such as pain, fatigue and weakness.
* Functional limitations and disabilities, such as loss of independence in activities of daily living (e.g., grooming, bathing, dressing, driving a car), work and social and recreational activities.

It will identify factors associated with these problems and try to determine their relationship to them.

Patients 18 years of age and older with stage I, II, III or IV breast cancer may be eligible for this study. Participants will be drawn from patients referred to the National Naval Medical Center for diagnosis and treatment during 2000-20001.

Participants will be interviewed and their medical records reviewed for past medical history, history of the present illness and social and recreational history. They will be seen five times over a 1-year period (initial visit and at 3, 6, 9, and 12 months), for 30-minute visits, which will include the following:

* Interview about past medical history and present illness, social and recreational activities, functional independence at work and during activities of daily living.
* Complete health survey and upper limb disability questionnaire; physical activity questionnaire to be completed at 6 and 12 months after medical treatment begins. The questionnaires take about 30 to 40 minutes to complete.
* Upper body examination, including pain measurement using a 10-point scale, an upper limb lift test, and measures of upper limb volume and girth.

DETAILED DESCRIPTION:
This retrospective (case-control) outcome study will investigate the frequency and severity of morbidities in a population of approximately 160 patients diagnosed with breast cancer before and after medical and surgical treatment. Subjects will be followed for one-year with quarterly examinations (baseline [pre-medical treatment] and at 1, 3 months, 6 months, 9 months and 12 months after treatment). In order for cancer survivors to understand the risk of impairment and functional limitations, and disability; and for health care providers to determine the risk of physical impairment, functional limitations, and loss of independence (morbidity) in patients with breast cancer; it is necessary to study these patients from the point of diagnosis (before surgery) to a reasonable period following the completion of the primary treatment program (1 year after medical treatment). Although pain, numbness, fatigue, lymphedema and diminished physical function are described as prevalent and debilitating conditions, remarkably few clinical studies are published describing the associated physical impairments, functional limitations or on methods for their control with measures prior to medical intervention and long-term follow-up. While several past reports have identified the impact of medical and surgical intervention on symptom distress and functional capacity of these patients, these studies do not provide sufficient evidence to identify the: 1) level of physical impairment that predicts morbidity in these patients, 2) individual factors that are specific predictors of morbidity in these patients, or 3) time period in which these morbidities occur. The majority of previous studies investigating morbidity of patients with breast cancer following medical and surgical intervention are cross-sectional, case series, retrospective analysis without a comparison/control group and without baseline measures prior to intervention. The proposed outcome study will include: 1) a retrospective review of specific medical record information such as staging conference information and the standard clinical quarterly examination during a one year period, and 2) administration of a follow-up outcome questionnaire, a physical activity questionnaire and a quality of life questionnaire at the 6 and 12 months time points. The outcome survey is an upper limb disability questionnaire developed as an outcome measure for this project. Data available in these measurement domains will allow the researchers to determine the: 1) frequency and severity of: a) symptom distress (fatigue, pain including chronic pain, aching, weakness, burning, tingling, numbness, anxiety, and depression) and pathological conditions (adhesive capsulitis, weakness and atrophy, neuropathy, scar/skin adhesions, lymphedema), b) physical impairments (diminished upper extremity and trunk range of motion/flexibility, strength, coordination and increased girth), and c) functional imitations and disabilities during the course of the medical treatment (loss of independence in or ability to perform routine activities of daily living i.e., grooming, bathing, dressing, driving an automobile, and in some cases, return to their regular work, recreational and social activities). 2) level of impairment at which these patients have lost independence in function and identity those patients at higher risk for the loss of independence in function (e.g., ADL's).

ELIGIBILITY:
* INCLUSION CRITERIA:

Population/Subjects: Individuals with breast cancer are identified among the patient population at National Naval Medical Center (NNMC). Patients referred to the NNMC Breast Care Center (NNMC-BCC) for diagnosis and management (surgical treatment and radiation treatment or chemotherapy) of histologically established breast cancer (stage I, II, III, or IV) during 2000-2001, are eligible to participate in the study.

Subjects must be over age 18. This age ensures they are post-puberty as breast cancer does not occur prior to puberty; and been seen pre-surgical or medical intervention for baseline measurements and agree to participate in five follow-up visits of 30 minutes in duration during the next year.

EXCLUSION CRITERIA:

Subject's medical records are unavailable and clinical examination forms are incomplete.

Subjects choose not to participate in the study.

Subjects are unable to complete the questionnaires.

Subjects are under age 18.

Men are not excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2001-11-16; Study Completion 2016-08-17

PRIMARY OUTCOMES:
Upper limb strength | 1,3,6,9,12,60 months
Range of motion | 1,3,6,9,12,60 month
Upper limb volume | 1,3,6,9,12,60 month

CONTACTS AND LOCATIONS:
Overall Officials: Minal Jain, R.P.T., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] King KB, Nail LM, Kreamer K, Strohl RA, Johnson JE. Patients' descriptions of the experience of receiving radiation therapy. Oncol Nurs Forum. 1985 Jul-Aug;12(4):55-61. No abstract available. PMID 3847996
- [Background] Meyerowitz BE, Watkins IK, Sparks FC. Quality of life for breast cancer patients receiving adjuvant chemotherapy. Am J Nurs. 1983 Feb;83(2):232-5. No abstract available. PMID 6549885
- [Background] Carter BJ. Women's experiences of lymphedema. Oncol Nurs Forum. 1997 Jun;24(5):875-82. PMID 9201739